CLINICAL TRIAL: NCT06439810
Title: Diagnostic Utility of Mycobacterium Tuberculosis Cell-free DNA (MTB cfDNA) in Tuberculous and Non-tuberculous Pleural Effusion
Brief Title: Diagnostic Utility of Mycobacterium Tuberculosis Cell-free DNA
Acronym: MYDNITE
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Doctor (Assistant Professor), Chinese University of Hong Kong
Other Study IDs: PF_MTB cfDNA
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Tuberculosis, Pleural
Keywords: Tuberculosis; Tuberculous pleuritis; cell-free DNA
MeSH Terms: conditions — Tuberculosis, Pleural; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pleural fluid for cell-free DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tuberculous pleuritis: Patients with definite or probable tuberculous pleuritis
  Interventions: Diagnostic Test: Mycobacterium tuberculosis (MTB) cell-free DNA (cfDNA)
- Non-tuberculous pleuritis: Patients without tuberculous pleuritis
  Interventions: Diagnostic Test: Mycobacterium tuberculosis (MTB) cell-free DNA (cfDNA)

INTERVENTIONS:
Diagnostic Test: Mycobacterium tuberculosis (MTB) cell-free DNA (cfDNA) — Comparing the diagnostic accuracy between MTB cfDNA and PCR on diagnosing tuberculous pleuritis
  Other Names: Mycobacterium tuberculosis PCR

SUMMARY:
Tuberculosis (TB) is one of the major global health threats and is the second leading infectious cause of death after COVID-19 in 2022. Extrapulmonary TB (EPTB), amongst which tuberculous pleuritis (TBP) is one of the most common subtypes, poses additional obstacles to global TB control due to its difficulty in diagnosis.

The diagnosis of TBP is challenging. The ideal way of confirming TBP is by direct detection of TB bacteria or its specific component in the pleural space. However, the performance of available diagnostic tests is far from satisfactory, and no single test can achieve multiple diagnostic goals simultaneously, including high detection sensitivity, high specificity to exclude other diseases, low invasiveness and detection of drug resistance. The inability to diagnose TBP early leads to unnecessary invasive pleural procedures and delayed curative treatment. There is a pressing need for a better diagnostic test to diagnose TBP confidently.

When TB bacteria die or break down, the DNA materials shed into the pleural space, forming Mycobacterium tuberculosis cell-free DNA (MTB cfDNA), which may aid in diagnosing TBP. However, only limited literature explored this aspect, and the sensitivity rates reported were still suboptimal due to the scarcity of DNA materials in the pleural fluid. Based on a small patient cohort, our group has recently developed a new laboratory assay measuring MTB cfDNA to overcome this problem, with a superior diagnostic performance to conventional tests. This assay can potentially capture the genes harbouring drug resistance towards anti-TB medications.

There are three aims in this research proposal. First, the diagnostic accuracy of the new MTB cfDNA assay in diagnosing TBP will be determined using a large cohort containing pleural fluid samples of various causes from countries with different TB burdens. Second, the clinical and laboratory factors determining the pleural fluid MTB cfDNA level will be identified. Third, the ability of the assay to capture different anti-TB drug-resistance genes will be explored.

This new diagnostic method will significantly enhance the pickup rate of TBP, benefit patients with less invasive procedures, shorter hospital stays and timely treatment.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a key infectious disease burden globally. According to the Global TB Report by the World Health Organization (WHO) in 2023, TB is the second leading infectious cause of death after COVID-19 in 2022. Extrapulmonary TB, amongst which tuberculous pleuritis (TBP) is one of the most common subtypes, poses additional obstacles to global TB control due to its difficulty in diagnosis. There is a large geographical variation in the incidence of TBP, with the proportion of TBP among all TB patients ranging from 2.2% to 31.4%. An increasing incidence of TBP was noted in two large retrospective Chinese cohort studies.

The paucibacillary nature of TBP leads to its diagnostic challenge. Despite being a gold standard diagnostic test, the diagnostic sensitivity of pleural fluid Mycobacterium tuberculosis (MTB) culture is suboptimal. It varies between 7.0% and 75.0%, depending on the culture medium and HIV status. Its long turnaround time of around 4 to 8 weeks also impairs its clinical practicality. Commercial PCR techniques, such as Xpert MTB/RIF or Xpert Ultra, are rapid and specific tests with positive results. However, their utilities are limited by suboptimal sensitivity. Pleural biopsy for histology and combined histology / culture might raise the sensitivity to 66% and 79%, but this procedure is more invasive than thoracentesis. Pleural fluid adenosine deaminase (ADA) is the most commonly studied biomarker, with diagnostic sensitivity and specificity of 0.93 and 0.90 at a cutoff of 40 U/L. Its cutoff range may vary with patient characteristics (age, comorbid illness). The difficulty in diagnosing TBP, therefore, leads to delayed initiation of anti-TB treatment. Empirical anti-TB treatment may be initiated based on compatible clinical presentations without confirmatory diagnostic microbiological results, bearing the risk of treatment toxicities (e.g. hepatotoxicity). This suggests an unmet clinical need for a better diagnostic tool for TBP.

Detecting MTB cell-free DNA (cfDNA) in the pleural fluid may solve the above problems. It is a potential diagnostic tool with minimal invasiveness and, most importantly, a direct confirmation of MTB in the pleural space. However, previous PCR-based methods reported suboptimal sensitivity for diagnosing TBP, of about 40-80%. The sensitivity may be limited by the low level of MTB cfDNA and the single-gene target (IS6110 or devR) in the detection. With the advancement of next-generation sequencing (NGS) technology, the detection of microbial cfDNA by metagenomic NGS (mNGS) has been applied in infectious disease diagnostics. Chang et al. have previously evaluated the use of mNGS in blood and urine samples for tuberculosis diagnostics. They revealed that such methodology is limited by the low MTB concentration and the background of contaminating non-tuberculous mycobacterial (NTM) DNA, which shares similar sequences to the pathogenic MTB.

Our group has recently developed a new laboratory assay measuring the MTB cfDNA levels. We hypothesise that the new MTB cfDNA assay has better diagnostic performance than conventional microbiological methods in discriminating pleural effusions due to TBP from non-TBP. Since the development cohort only contains a limited number of pleural fluid samples, a large-scale confirmatory study containing pleural effusions with a wide spectrum of causes is required to confirm its clinical utility before being introduced in clinical practice. This study has three major aims. First, the diagnostic accuracy of the new MTB cfDNA assay in diagnosing TBP will be determined using a large cohort containing pleural fluid samples of various causes from countries with different TB burdens. Second, the clinical and laboratory factors determining the pleural fluid MTB cfDNA level will be identified. Third, the ability of the assay to capture different anti-TB drug-resistance genes will be explored on pleural fluid from DR-TB endemic areas.

ELIGIBILITY:
Inclusion Criteria:

* New-onset pleural effusion planning for thoracentesis
* Age 18 years or above
* Able to give informed consent

Exclusion Criteria:

* History of TBP or intrapleural therapy (including talc and fibrinolytic) in the ipsilateral pleural space. Patients with a history of TB outside the pleural space completed anti-TB treatment can be included
* History of surgical intervention (including decortication, pleurodesis, lung resection) in the ipsilateral pleural space
* Concomitant use of at least two anti-TB medications (including isoniazid, rifampicin, pyrazinamide, ethambutol, amikacin, streptomycin, levofloxacin, moxifloxacin, linezolid) for more than consecutive 7 days in the past 3 months
* Consent not obtained from the participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with definite or probably TBP will be recruited as positive control. Patients without TBP will be recruited as negative control
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of the new MTB cfDNA assay | 24 months
  to evaluate the diagnostic accuracy of the new MTB cfDNA assay in a randomly selected cohort of pleural effusions containing TBP and non-TBP aetiologies.

SECONDARY OUTCOMES:
Diagnostic performance of the new MTB cfDNA assay | 24 months
  Diagnostic performance of the new MTB cfDNA assay with MTB PCR in diagnosing MTB culture-positive and MTB culture-negative TBP
Clinical factors that may affect the levels of MTB cfDNA in TBP | 24 months
  Clinical and laboratory factors may affect MTB cfDNA levels in pleural fluid
Diagnostic performance of the new MTB cfDNA assay (drug resistant TB) | 24 months
  Diagnostic performance of the new MTB cfDNA assay in capturing drug resistance genes towards anti-TB medications

CONTACTS AND LOCATIONS:
Overall Officials: Ka Pang Chan, MBChB, Principal Investigator — Prince of Wales Hospital

IPD SHARING:
Plan to Share IPD: No